CLINICAL TRIAL: NCT05295940
Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3841136 in Healthy and Overweight Participants
Brief Title: A Study of LY3841136 in Healthy and Overweight Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18309; J3R-MC-YDAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-03-24; First posted 2022-03-25 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Healthy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3841136 (Part A) (Experimental): Single ascending doses of LY3841136 administered subcutaneously (SC).
  Interventions: Drug: LY3841136
- LY3841136 (Part B) (Experimental): Multiple ascending doses of LY3841136 administered SC.
  Interventions: Drug: LY3841136
- Placebo (Part A) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3841136 — Administered SC.
  Arms: LY3841136 (Part A); LY3841136 (Part B)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3841136 in healthy and overweight participants. Blood tests will be performed to check how much LY3841136 gets into the bloodstream and how long it takes the body to eliminate it. This is a 2-part study and may last up to 14 and 28 weeks for each participant and may include 7 and 19 visits in parts A and B, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who agree to use highly effective/effective methods of contraception and female participants not of childbearing potential
* Have had a stable weight for the last 3 months
* Have a body mass index (BMI) in the range of 18.5 to 32 kilogram per square meter (kg/m²), both inclusive (in Part A) or a BMI in the range of 27 to 40 kg/m², both inclusive (in Part B)

Exclusion Criteria:

* Are women who are lactating
* Have known allergies to related compounds of LY3841136 or any components of the formulation
* Have a history of significant atopy (severe or multiple allergic manifestations), or clinically significant multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions
* Have been diagnosed with Type 1 or Type 2 diabetes mellitus
* Have a history of chronic medical conditions involving the heart, liver, or kidneys

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Predose up to 14 weeks (Part A) & 28 weeks (Part B)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3841136 | Predose through week 14 (Part A) & week 28 (Part B)
  PK: AUC of LY3841136
PK: Maximum Observed Concentration (Cmax) of LY3841136 | Predose through week 14 (Part A) & week 28 (Part B)
  PK: Cmax of LY3841136
Pharmacodynamics (PD): Change From Baseline in Body Weight | Predose through week 28
  PD: Change From Baseline in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Briere DA, Qu H, Lansu K, He MM, Moyers JS, Coskun T, Long A, Allen D, O'Farrell L, Bowen B, Pratt E, Tidemann-Miller B, Tham LS, Ibriga H, Alsina-Fernandez J, Mather KJ, Haupt A, Bhattachar SN. Eloralintide (LY3841136), a novel amylin receptor agonist for the treatment of obesity: From discovery to clinical proof of concept. Mol Metab. 2025 Dec;102:102271. doi: 10.1016/j.molmet.2025.102271. Epub 2025 Oct 16. PMID 41109426